CLINICAL TRIAL: NCT01084213
Title: A Trial of Intermittent Preventive Treatment With Sulfadoxine-pyrimethamine Versus Intermittent Screening and Treatment of Malaria in Pregnancy
Brief Title: Intermittent Preventive Treatment Versus Scheduled Screening and Treatment of Malaria in Pregnancy
Acronym: IPTp_IST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research and Training Centre, Mali (Unknown); University of Ouagadougou, Burkina Faso (Other); Medical Research Council Unit, The Gambia (Other); Navrongo Health Research Centre, Ghana (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MiPcMA05
Record Dates: First submitted 2010-03-03; First posted 2010-03-10 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Malaria; Pregnancy; Anaemia
Keywords: Low birth weight; Placenta malaria; Anaemia; Intermittent preventive treatment; Intermittent screening and treatment; Rapid diagnostic test
MeSH Terms: conditions — Malaria; Anemia | interventions — Pregnancy; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPTp with SP (Active Comparator): Study women will receive at least two doses of SP during their pregnancy, one at each of the recommended ante-natal visits during the 2nd and 3rd trimester.
  Interventions: Drug: SP-IPTp
- IST using RDTs (Experimental): Scheduled intermittent screening using rapid diagnostic tests and treatment of those who are RDT positive during ante-natal clinic visits in the 2nd and 3rd trimester.
  Interventions: Drug: Intermittent screening and treatment of malaria in pregnancy (IST)

INTERVENTIONS:
Drug: Intermittent screening and treatment of malaria in pregnancy (IST) — Scheduled intermittent screening of study women using rapid diagnostic test and treatment of those who are RDT positive during ante-natal clinic visits in the 2nd and 3rd trimester with arthemether lumefantrine.
  Other Names: Coartem
  Arms: IST using RDTs
Drug: SP-IPTp — Study women will receive at least two doses of Sulfadoxine Pyrimethamine during their pregnancy, one at each of the recommended ante-natal visits during the 2nd and 3rd trimester.
  Other Names: SP
  Arms: IPTp with SP

SUMMARY:
The incidence of malaria, including the incidence in pregnant women, is declining in many African countries. Thus, there is a need to re-examine the efficacy and cost effectiveness of giving intermittent preventive treatment with sulphadoxine-pyrimethamine in pregnancy (SP-IPTp) on several occasions during pregnancy, an intervention that is threatened by increasing resistance to SP. Possible alternatives to SP-IPTp need to be explored. This applies especially to areas with highly seasonal malaria transmission where women are at risk for only a short period of the year.

The goal of this project is to determine whether in pregnant women who sleep under a long lasting insecticide treated bed net, screening and treatment at each scheduled antenatal clinic visit is as effective in protecting them from anaemia, low birth weight and placental infection as SP-IPTp.

Primigravidae and secundigravidae who present at antenatal clinics in study sites in four West African countries (Burkina Faso, Ghana, Mali and The Gambia) will be randomised to one of two groups. All women will be given a long lasting insecticide treated bed net on first presentation at the antenatal clinic. Women in group 1 (reference group) will receive SP-IPTp according to the current WHO guidelines. Those in group 2 will be screened with a rapid diagnostic test at each scheduled antenatal clinic visit and treated if parasitaemic. Approximately 5000 women will be recruited, 2500 in each group. Women will be encouraged to deliver in hospital where maternal haemoglobin and birth weight will be recorded and a placental sample obtained. Those who deliver at home will be visited within a week of delivery and maternal haemoglobin and infant weight recorded. Mothers and infants will be seen again six weeks after delivery. Also at delivery peripheral maternal blood sample will be obtained for the diagnosis of malaria using RDT, microscopy and PCR. The primary end points of the trial will be birth weight and anaemia at 38 weeks (+/-2 weeks) of gestation. The study is powered to show non-inferiority of group 2 compared to group 1. The costs and cost effectiveness of each intervention will be evaluated.

In the light of recent evidence suggesting that malaria infection during pregnancy, particularly in the last trimester may influence an infant's risk of malaria, we proposed to follow infants born to mothers recruited in the Navrongo site in Ghana who have received either IST or IPTp in pregnancy throughout the whole of their first year of life beyond the six weeks originally proposed. We have received approval for this from the ethic committees at Kwame Nkrumah University of Science and Technology, Ghana Health Service and Navrongo Health Research Centre. The aim is to obtain information on the incidence of both symptomatic and asymptomatic malaria infections in these infants during follow up of the infants.

The study will provide information to national malaria control programmes on whether there are alternative, safe and effective methods to the SP IPTp regimen for reducing the burden of malaria in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a first or second pregnancy.
2. Gestation between 16 to 30 weeks inclusive at first booking as determined by symphysio-fundal measurements.
3. Provision of informed consent to join the trial.
4. Residence in the study area and intention to stay in the area for the duration of the pregnancy.

Exclusion Criteria:

1. Absence of informed consent.
2. An intention to leave the study area before delivery.
3. A history of sensitivity to sulphonamides.
4. Clinical AIDS or known HIV positivity.
5. Presence of any systemic illness likely to interfere with interpretation of the results of the trial.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5354 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of low birth weight | 6 - 18 months
Prevalence of third trimester anaemia | 3 - 12 months
Prevalence of placenta malaria | 6 - 18 months

SECONDARY OUTCOMES:
Prevalence of anaemia at the time of delivery or shortly afterwards. | 6 - 18 months
Prevalence of peripheral blood parasitaemia | 6 - 18 months
Episodes of clinical malaria during the course of the pregnancy. | 1 year
Serious adverse events in the mother. | 6 - 18 months
Adverse outcome of pregnancy - abortions, still births and neonatal deaths. | 6 - 18 months
Occurrence of congenital abnormalities. | 6 - 18 months
Feasibility and costs of each approach to the control of malaria in pregnancy. | 1 year
Cost per cases of maternal anaemia (severe and non-severe) and peripheral malaria averted. | 1 year
Acceptability of each approach by pregnant women and antenatal clinic staff. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Greenwood, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Paul Milligan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Feiko T Kuile, PhD, Principal Investigator — Liverpool School of Tropical Medicine, UK; Harry Tagbor, DrPH, Principal Investigator — Kwame Nkrumah University of Science & Technology, School of Medical Sciences, Ghana
Locations (4):
- Université de Ouagadougou, Ouagadougou, Burkina Faso
- Navrongo Health Research Centre, Navrongo, Ghana
- Medical Research and Training Centre, Bamako, Mali
- Medical Research Council Laboratories, Basse Santa Su, The Gambia

REFERENCES:
- [Derived] Berry I, Walker P, Tagbor H, Bojang K, Coulibaly SO, Kayentao K, Williams J, Oduro A, Milligan P, Chandramohan D, Greenwood B, Cairns M. Seasonal Dynamics of Malaria in Pregnancy in West Africa: Evidence for Carriage of Infections Acquired Before Pregnancy Until First Contact with Antenatal Care. Am J Trop Med Hyg. 2018 Feb;98(2):534-542. doi: 10.4269/ajtmh.17-0620. Epub 2017 Nov 30. PMID 29210351
- [Derived] Tagbor H, Cairns M, Bojang K, Coulibaly SO, Kayentao K, Williams J, Abubakar I, Akor F, Mohammed K, Bationo R, Dabira E, Soulama A, Djimde M, Guirou E, Awine T, Quaye S, Njie F, Ordi J, Doumbo O, Hodgson A, Oduro A, Meshnick S, Taylor S, Magnussen P, ter Kuile F, Woukeu A, Milligan P, Chandramohan D, Greenwood B. A Non-Inferiority, Individually Randomized Trial of Intermittent Screening and Treatment versus Intermittent Preventive Treatment in the Control of Malaria in Pregnancy. PLoS One. 2015 Aug 10;10(8):e0132247. doi: 10.1371/journal.pone.0132247. eCollection 2015. PMID 26258474